CLINICAL TRIAL: NCT00498615
Title: Efficacy, Tolerability and Biology of a Rho-kinase Inhibitor (Fasudil) in the Treatment of Raynaud's Phenomenon
Brief Title: A Rho-kinase Inhibitor (Fasudil) in the Treatment of Raynaud's Phenomenon
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Fredrick M. Wigley, Professor of Medicine, Johns Hopkins University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00002801
Record Dates: First submitted 2007-07-06; First posted 2007-07-10 (Estimated); Results first posted 2014-11-04 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-08

CONDITIONS: Raynaud; Scleroderma
Keywords: scleroderma; Raynaud's phenomenon; Rho-kinase inhibitor
MeSH Terms: conditions — Scleroderma, Diffuse; Raynaud Disease | interventions — fasudil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fasudil 80 mg (Experimental): Subject is given a single dose of 80 mg of Fasudil ( blinded to participant and researcher) a cold challenge is given 2 hrs after the dose.
  Interventions: Drug: Fasudil
- 40 mg Fasudil (Experimental): Subject is given a single dose of 40 mg of Fasudil ( blinded to participant and researcher) a cold challenge is given 2 hrs after the dose.
  Interventions: Drug: Fasudil
- placebo (Placebo Comparator): Subject is given a single dose of placebo( blinded to participant and researcher) a cold challenge is given 2 hrs after the dose.
  Interventions: Drug: Fasudil

INTERVENTIONS:
Drug: Fasudil — Each subject will be randomly assigned to 1 of 6 possible treatment sequences (ABC, ACB, BAC, BCA, CAB, and CBA) in a double-blind manner: A- a single oral dose of 2 placebo tablets; B- a single, oral 40 mg Fasudil dose as one 40 mg tablet and 1 placebo tablet; C- a single oral 80 mg dose as two 40 mg Fasudil tablets. Subjects will be randomized at the screening/baseline visit to a specific treatment sequence based upon a computer generated code on a 1:1:1:1:1:1 ratio for the 6 possible sequences. A single dose consisting of the two tablets will be taken after fasting for 10 hours once during each treatment period. A washout interval of at least 24 hours and no more than 7 days will be maintained between treatment periods. Concomitant medications will not be taken during the study session.
  Other Names: No other name found

SUMMARY:
Raynaud's phenomenon is thought to occur when, in response to cold or emotional stress, there is closure of the digital arteries and cutaneous arterioles leading to the clinical finding of sharp demarcated digital pallor and cyanosis of the distal skin of the fingers and/or toes. Patients often continue to experience problems despite current available treatment. The investigators' study will investigate the use of a new vasodilator called Fasudil, a Rho-kinase inhibitor. The investigators' hypothesis is that Fasudil will prevent vasoconstriction of digital and cutaneous arteries during a standard laboratory based cold exposure and will therefore improve digital blood flow and skin temperature recovery time following cold challenge. These data will provide the rationale for a more elaborate clinical trials in real life situations.

DETAILED DESCRIPTION:
Raynaud's phenomenon (RP) is a reversible vasospastic disorder of digital arteries and cutaneous arterioles characterized by typical skin color changes and tissue ischemia (1). Avoidance of common triggers such as cold temperatures and emotional stress often leads to improvement of symptoms. When such a strategy yields inadequate benefits, pharmacologic therapy is needed.

Cutaneous vasoconstriction occurs through a general sympathetic adrenergic response and through local mechanisms in response to cold. While under normal conditions, the vasomotor tone is regulated mainly by a.2A- adrenoreceptors (a.2A-AR) expressed on vascular smooth muscle cells (VSMC) (2); during cold exposure the normally "silent" a.2C-AR relocate from the Golgi complex to the cell surface, driving the cold-induced vasoconstrictive response (3). Interestingly, the reactivity to a.2-AR stimulation is highly increased in cutaneous arteries of patients with systemic sclerosis (SSc; scleroderma) (4), and block- age of a.2C-AR has shown to shorten the time to recover digital skin temperature after a cold challenge in patients with Raynaud's Phenomenon secondary to Scleroderma (5).

The RhoA/Rho kinase pathway is activated by cooling and mediates vasoconstriction of cutaneous arteries by inducing a.2C-AR relocation to the cell surface and by increasing calcium-dependent Vascular Smooth Muscle Cells (VSMC )contractility (6). Rho kinase inhibition has been shown to effectively reduce

a.2-AR-mediated response during cold exposure and to prevent cold-induced vasoconstriction in human skin (6) Therefore, RhoA/Rho kinase inhibition may provide a highly selective intervention directed toward the mechanisms underlying thermosensitive vasomotor responses in the skin of Raynaud's Phenomenon patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of scleroderma
* definite Raynaud's

Exclusion Criteria:

* symptomatic orthostatic hypotension
* evidence of current malignancy
* active ischemic digital ulcer and/or tissue gangrene
* history of sympathectomy at any time
* upper extremity deep vein thrombosis or lymphedema within 3 months of the study
* recent surgical procedure requiring general anesthesia
* current alcohol or illicit drug use
* use of any investigational drug within 30 days of the study sessions
* pregnancy or current breast feeding
* subjects felt by the investigators to active disease that would affect their ability to safely participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fredrick M Wigley, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Subjects received a single dose of Fasudil 80 mg at treatment period 1. At treatment period 2 they will received a single dose of Fasudil 40 mg and at treatment period 3 they received a single dose of placebo. A washout interval of at least 24 hours and no more than 7 days will be maintained between treatment periods.
- Sequence 2: Subjects received a single dose of Fasudil 40 mg at treatment period 1. At treatment period 2 they will received a single dose of Fasudil 80 mg and at treatment period 3 they received a single dose of placebo. A washout interval of at least 24 hours and no more than 7 days will be maintained between treatment periods
- Sequence 3: Subjects received a single dose of Fasudil 80 mg at treatment period 1. At treatment period 2 they will received a single dose of placebo and at treatment period 3 they received a single dose of Fasudil 40 mg. A washout interval of at least 24 hours and no more than 7 days will be maintained between treatment periods
- Sequence 4: Subjects received a single dose of placebo at treatment period 1. At treatment period 2 they will received a single dose of Fasudil 40 mg and at treatment period 3 they received a single dose of Fasudil 80 mg. A washout interval of at least 24 hours and no more than 7 days will be maintained between treatment periods
- Sequence 5: Subjects received a single dose of Fasudil 40 mg at treatment period 1. At treatment period 2 they will received a single dose of placebo and at treatment period 3 they received a single dose of Fasudil 80 mg. A washout interval of at least 24 hours and no more than 7 days will be maintained between treatment periods
- Sequence 6: Subjects received a single dose of placebo at treatment period 1. At treatment period 2 they will received a single dose of Fasudil 80 mg and at treatment period 3 they received a single dose of Fasudil 40 mg. A washout interval of at least 24 hours and no more than 7 days will be maintained between treatment periods
Period: Fasudil 80mg
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 2 | 4 | 3 | 2 | 3 | 3
Completed | 2 | 4 | 3 | 2 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Fasudil 40mg
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 2 | 4 | 3 | 2 | 3 | 3
Completed | 2 | 4 | 3 | 2 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Placebo
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 2 | 4 | 3 | 2 | 3 | 3
Completed | 2 | 4 | 3 | 2 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Men and women between ages 18-80 years with a clinical diagnosis of Raynauds Phenomenon secondary to Scleroderma were eligible for the study.
Groups:
- 3 Period Crossover Study ( All Participants): This is a single-center, double-blind, placebo-controlled, randomized, 3-period crossover study of oral fasudil (40 mg or 80 mg) or placebo administered 2 hours before a standardized cold challenge.
  Men and women between ages 18-80 years with a clinical diagnosis of RP secondary to SSc were eligible for the study.
Arm/Group | 3 Period Crossover Study ( All Participants)
Number analyzed (Participants) | 17
Age, Continuous [Mean (Full Range); unit: years] | 51 [30 to 70]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: The Time to Recover 50% of Fall in the Baseline Skin Temperature.
Description: The time to recover 50% of the drop from baseline (prechallenge) skin temperature was derived for each subject for each cold challenge. After each of 3 study interventions received by each participant. Each participant received Fasudil 4o mg, 80 mg and placebo in a randomized sequence blinded to the participant and researchers.
Time Frame: within 60 minutes
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- 40 mg Fasudil: This is a single-center, double-blind, placebo-controlled, randomized, 3-period crossover study of oral fasudil 40 mg administered 2 hours before a standardized cold challenge participant and researchers will not know what is received on the testing day.
- 80 mg Fasudil: participants will receive 80mg of Fasudil at 1 one 3 study periods 2hrs before a cold challenge.
- Placebo: participants will receive placebo at 1 of 3 study periods. participants and researchers will not know which is received.
Arm/Group | 40 mg Fasudil | 80 mg Fasudil | Placebo
Number analyzed (Participants) | 17 | 17 | 17
minutes | 7.5 (3.2) | 8.2 (3.0) | 7.9 (3.1)

2. Secondary Outcome: The Blood Flow by Laser Doppler Scans of the Fingers
Description: The measurement of the blood flow of participants prior to cold challenge 2 hours after receiving study.
Time Frame: Blood flow prior to cold challenge 2 hours after taking study drug
Measure: Mean (Standard Deviation); unit: perfusion units
Groups:
- 80 mg Fasudil: This is a single-center, double-blind, placebo-controlled, randomized, 3-period crossover study of oral fasudil In this arm participants received 80 mg of Fasudil 2 hours before a standardized cold challenge.
  Men and women between ages 18-80 years with a clinical diagnosis of Raynauds Phenomenon secondary to Scleroderma were eligible for the study.
- 40 mg Fasudil: In this group participants received 40mg of Fasudil 2 hours before cold challenge
- Placebo: In this group participants received placebo 2 hours before cold challenge.
Arm/Group | 80 mg Fasudil | 40 mg Fasudil | Placebo
Number analyzed (Participants) | 17 | 17 | 17
perfusion units | 138.3 (55.1) | 134.1 (73.4) | 122.6 (57.6)

3. Primary Outcome: Time to Recover to 70% of Fall in the Baseline Skin Temperature After Cold Challenge.
Description: The time to recover 70% of the drop from baseline (prechallenge) skin temperature was derived for each subject for each cold challenge. After each of 3 study interventions received by each participant. Each participant received Fasudil 4o mg, 80 mg and placebo in a randomized sequence blinded to the participant and researchers.
Time Frame: within 60 minutes
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Fasudil 80 mg: Time to recover 70% of baseline skin temperature after cold challenge done 2 hrs after dose.
  Fasudil: Each subject will be randomly assigned to 1 of 6 possible treatment sequences (ABC, ACB, BAC, BCA, CAB, and CBA) in a double-blind manner: A- a single oral dose of 2 placebo tablets; B- a single, oral 40 mg Fasudil dose as one 40 mg tablet and 1 placebo tablet; C- a single oral 80 mg dose as two 40 mg Fasudil tablets. Subjects will be randomized at the screening/baseline visit to a specific treatment sequence based upon a computer generated code on a 1:1:1:1:1:1 ratio for the 6 possible treatments. A single dose consisting of the two tablets will be taken after fasting for 10 hours once during each treatment period. A washout interval of at least 72 hours and no more than 7 days will be maintained between treatment periods. Concomitant medications will not be taken during the study session.
- 40 mg Fasudil: Time to reach 70% skin temperature after cold challenge done 2 hrs after dosing.
  Fasudil: Each subject will be randomly assigned to 1 of 6 possible treatment sequences (ABC, ACB, BAC, BCA, CAB, and CBA) in a double-blind manner: A- a single oral dose of 2 placebo tablets; B- a single, oral 40 mg Fasudil dose as one 40 mg tablet and 1 placebo tablet; C- a single oral 80 mg dose as two 40 mg Fasudil tablets. Subjects will be randomized at the screening/baseline visit to a specific treatment sequence based upon a computer generated code on a 1:1:1:1:1:1 ratio for the 6 possible treatments. A single dose consisting of the two tablets will be taken after fasting for 10 hours once during each treatment period. A washout interval of at least 72 hours and no more than 7 days will be maintained between treatment periods. Concomitant medications will not be taken during the study session.
- Placebo: Time to reach 70% of skin temperature after cold challenge done 2 hrs after taking placebo
  Fasudil: Each subject will be randomly assigned to 1 of 6 possible treatment sequences (ABC, ACB, BAC, BCA, CAB, and CBA) in a double-blind manner: A- a single oral dose of 2 placebo tablets; B- a single, oral 40 mg Fasudil dose as one 40 mg tablet and 1 placebo tablet; C- a single oral 80 mg dose as two 40 mg Fasudil tablets. Subjects will be randomized at the screening/baseline visit to a specific treatment sequence based upon a computer generated code on a 1:1:1:1:1:1 ratio for the 6 possible treatments. A single dose consisting of the two tablets will be taken after fasting for 10 hours once during each treatment period. A washout interval of at least 72 hours and no more than 7 days will be maintained between treatment periods. Concomitant medications will not be taken during the study session.
Arm/Group | Fasudil 80 mg | 40 mg Fasudil | Placebo
Number analyzed (Participants) | 17 | 17 | 17
minutes | 17.1 (10.8) | 15.0 (9.4) | 18.2 (10.7)

ADVERSE EVENTS:
Time Frame: 35 days
Groups:
- Placebo: Placebo was administered 2 hours before a standardized cold challenge.
- 40 mg Fasudil: 40 mg Fasudil was administered 2 hours before a standardized cold challenge.
- 80mg Fasudil: 80mg Fasudil was administered 2 hours before a standardized cold challenge.
Arm/Group | Placebo | 40 mg Fasudil | 80mg Fasudil
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No